CLINICAL TRIAL: NCT05095844
Title: National Vaccine Adverse Event Reporting Survey to Determine the Etiology of Vaccine-Induced Injury
Brief Title: National Vaccine Adverse Event Reporting Survey and Etiology
Acronym: NVAERS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuroganics LLC (Industry)
Collaborators: Ramos Injury Law Firm (Unknown)
Responsible Party: Sponsor
Other Study IDs: NVAERS_1121
Record Dates: First submitted 2021-10-13; First posted 2021-10-27 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Vaccine Adverse Reaction; Vaccine Reaction; Vaccine or Biological Substance, Unspecified Causing Adverse Effects in Therapeutic Use; Corona Virus Infection; Blood Clot; Thrombocytopenia; Neuritis; Vasculitis; Influenza; Guillain-Barré; GWAS; Genetic Sequencing
Keywords: COVID-19; coronavirus; vaccine; influenza; injury; compensation; Pfizer; Moderna; BioNTech; Johnson and Johnson; Comirnaty; Flu Vaccination; Quadrivalent; Flucelvax; Flu Shots; Afluria Quadrivalent (Seqirus); Fluarix; FluLaval; Fluzone; Walgreens; CVS; Pharmacy
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Thrombosis; Thrombocytopenia; Neuritis; Vasculitis; Influenza, Human; Guillain-Barre Syndrome; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinated: All individuals who have received a vaccine dose.
  Interventions: Biological: vaccinated

INTERVENTIONS:
Biological: vaccinated — Pfizer-BioNTech COVID-19 Vaccine, Moderna or J&J/Janssen COVID-19 Vaccine, Diphtheria (e.g., DTP, DTaP, Tdap, DT, Td, TT) Haemophilus influenza type b polysaccharide conjugate vaccines (e.g., Hib) Hepatitis A (e.g., HAV) Hepatitis B (e.g., HBV) Human papillomavirus (e.g., HPV) Seasonal influenza (e.g., Flu) Measles (e.g., MMR) Mumps (e.g., MMR, MR, M) Meningococcal (e.g., MCV4, MPSV4, MenB-FHbp, MenB-4C) Pertussis (e.g., DTP, DTaP, Tdap) Pneumococcal conjugate (e.g., PCV) Polio (e.g., OPV or IPV) Rotavirus (e.g., RV) Rubella (e.g., MMR, MR, R) Tetanus (e.g., Td) Varicella (e.g., VAR)

SUMMARY:
If your serious vaccine-induced adverse event has been entered in the CDC Vaccine Adverse Event Reporting System (VAERS) we are interested in enrolling you for this study in order to log your symptoms.

The primary goal of this study is to create a national database and gather vaccine-associated serious adverse events/injury data from newly vaccinated individuals in the US in order to identify the possible underlying causal relationships and plausible underlying biological mechanisms. The project aims to identify the genetic determinants of vaccine-induced adverse response by studying host genetics. We plan to use whole genome sequencing to identify single nucleotide polymorphisms associated with cardiovascular, neurological, gastrointestinal, musculoskeletal and immunological symptoms induced by vaccine administration.

The secondary goal is to establish criteria that enable classification of vaccine-induced adverse events/injuries compare data from our database with the official Vaccine Injury Table National Vaccine Injury Compensation Program on or after March 21, 2017.

The tertiary goal is to establish a database to gather detailed long-term adverse reaction data from subjects enrolled in FDA Emergency Use Authorized vaccine clinical trials.

DETAILED DESCRIPTION:
Vaccinations are typically administered to healthy persons and often are mandated by states or federal authorities as a condition for school attendance or military service in order to prevent the spread of infectious diseases. Because vaccines are either mandated or recommended for vulnerable groups, such as children or the elderly, vaccines are often held to a higher standard of safety by the FDA than other medical products.

Due to the vast numbers of vaccine doses administered in the US there is a need to gather quality information on serious vaccine-associated adverse events leading to serious injury. Vaccine-induced adverse events are typically reported in the CDC Vaccine Adverse Event Reporting System (VAERS) database, which contains information on unverified reports of adverse events (illnesses, health problems and/or symptoms) following immunization with US-licensed vaccines. Reports are accepted from anyone and can be submitted electronically at www.vaers.hhs.gov.

The primary goal for this observational study is to establish an independent national database to classify vaccine-associated serious adverse events/injury data from vaccinated individuals. The plan is to gather survey data and health information from newly vaccinated individuals who have experienced serious adverse effects in order to help understand the possible causal relationships and plausible biological mechanisms underlying serious adverse events/injuries. The project aims to identify the genetic determinants of vaccine-induced adverse response by studying host genetics. We plan to use Nebula Genomics platform for whole genome sequencing to identify single nucleotide polymorphisms associated with cardiovascular, neurological, gastrointestinal, musculoskeletal and immunological symptoms induced by vaccine administration.

The secondary goal is to gather medical history and survey data from recently vaccinated individuals in order to develop a vaccine-injury risk assessment tool which may be used to predict individual vulnerability to vaccine adverse events/injury.

The tertiary goal is to establish a database to gather detailed long-term adverse reaction data from subjects enrolled in FDA Emergency Use Authorized vaccine clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Individuals who have received at least one vaccine dose of ANY of the following vaccines (below) and experienced adverse reaction within 60 days of vaccine administration:

1. Pfizer-BioNTech COVID-19 Vaccine
2. Moderna COVID-19 Vaccine
3. J&J/Janssen COVID-19 Vaccine
4. Diphtheria (e.g., DTP, DTaP, Tdap, DT, Td, TT)
5. Haemophilus influenza type b polysaccharide conjugate vaccines (e.g., Hib)
6. Hepatitis A (e.g., HAV)
7. Hepatitis B (e.g., HBV)
8. Human papillomavirus (e.g., HPV)
9. Seasonal influenza (e.g., Flu)
10. Measles (e.g., MMR)
11. Mumps (e.g., MMR, MR, M)
12. Meningococcal (e.g., MCV4, MPSV4, MenB-FHbp, MenB-4C)
13. Pertussis (e.g., DTP, DTaP, Tdap)
14. Pneumococcal conjugate (e.g., PCV)
15. Polio (e.g., OPV or IPV)
16. Rotavirus (e.g., RV)
17. Rubella (e.g., MMR, MR, R)
18. Tetanus (e.g., Td)
19. Varicella (e.g., VAR).

Exclusion Criteria:

1. Non citizens or permanent residents of the US
2. Individuals who have not received at least one vaccine dose in the past 3 years.
3. Individuals whose vaccine was administered more than 60 days before symptoms of the serious adverse event.

   -

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: US citizens or permanent residents and their dependents who have been vaccinated in the past 3 years and experienced a documented adverse event within 60 days of vaccination
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 2 years
  Reported adverse event occurring less than 60 days after administration of vaccine.

SECONDARY OUTCOMES:
Vaccine manufacturer efficacy | 2 years
  Comparison of multiple vaccine manufacturers for adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Cooper, Ph.D., Principal Investigator — Chief Science Officer/ Principal Investigator
Locations (1):
- Neuroganics LLC, Northglenn, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided